CLINICAL TRIAL: NCT02683018
Title: Investigation of Cannabis for Chronic Pain and Palliative Care
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: funding
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Diana Martinez, Research Scientist, New York State Psychiatric Institute
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 7220
Record Dates: First submitted 2016-02-11; First posted 2016-02-17 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smoked Cannabis High CBD/low THC (Active Comparator): Participants will visit the Marijuana Research Laboratory 3-5 weekdays per week for 4 weeks to be administered 1-2 Smoked Cannabis High CBD/low THC cigarettes (15.76% CBD; 3.11% THC) over the course of a 2-3 hour session.
  Interventions: Drug: Smoked Cannabis High CBD/low THC
- Smoked Placebo Cannabis Low CBD/low THC (Placebo Comparator): Participants will visit the Marijuana Research Laboratory 3-5 weekdays per week for 4 weeks to be administered 1-2 cannabis cigarettes (0.01% THC; 0.00% CBD) over the course of a 2-3 hour session.
  Interventions: Drug: Smoked Placebo Cannabis Low CBD/low THC

INTERVENTIONS:
Drug: Smoked Cannabis High CBD/low THC — Participants will visit the Marijuana Research Laboratory 3-5 weekdays per week for 4 weeks to be administered 1-2 cannabis cigarettes (15.76% CBD; 3.11% THC) over the course of a 2-3 hour session.
  Other Names: cannabis cigarettes (15.76% CBD; 3.11% THC)
  Arms: Smoked Cannabis High CBD/low THC
Drug: Smoked Placebo Cannabis Low CBD/low THC — Participants will visit the Marijuana Research Laboratory 3-5 weekdays per week for 4 weeks to be administered 1-2 cannabis cigarettes (0.01% THC; 0.00% CBD) over the course of a 2-3 hour session.
  Other Names: cannabis cigarettes (0.01% THC; 0.00% CBD)
  Arms: Smoked Placebo Cannabis Low CBD/low THC

SUMMARY:
The use of cannabis for severe medical conditions is being legalized in different states, increasing the mandate to make cannabis legal for medically ill patients. However, there is a lack of placebo-controlled studies investigating the efficacy of cannabis. Dronabinol (synthetic, oral Δ-9-THC) is FDA approved for the appetite stimulation in AIDS-related anorexia and nausea/vomiting in chemotherapy patients. Nabilone, a synthetic analogue of THC, is approved for nausea/vomiting in chemotherapy patients. These medications have been found to be effective for these disorders, but there remains an interest in studying cannabis, partly due to the numerous cannabinoids contained within the cannabis plant. Among these is cannabidiol, which does not produce subjective effects, but has been shown to have potent anti-inflammatory effects. In addition, there is data indicating that cannabidiol may be effective for neuropathic pain and nausea/vomiting.

The goal is to investigate the effects of high CBD/low THC cannabis on symptoms such as pain, nausea/vomiting, and quality of life in seriously ill participants. While there is data beginning to emerge that cannabis may have a beneficial effect on these symptoms, there are few placebo controlled, double-blind studies. Additionally, the administration of cannabis to medically ill patients may be limited by its subjective effects, such as anxiety, intoxication, or paranoia. Most cannabis available today has high levels of Δ-9-THC (about 15%). By using cannabis that is high in CBD, but low in - Δ-9-THC, it is hypothesized that some of these effects can be avoid, while maximizing the therapeutic effects, if any.

DETAILED DESCRIPTION:
The goal of this study is to perform a double-blind, placebo-controlled study to investigate the efficacy of cannabis, compared to placebo, in medically ill participants seeking relief symptoms such as pain, nausea, and vomiting. Participants who meet criteria for severe conditions will be referred from their clinicians . Cannabis that has a high concentration of cannabidiol, which is a cannabinoid that does not change perception or produce intoxication, and low in Δ-9-THC will be used. In this way, the hope is to maximize the benefit of cannabis, while lowering the possible side effects of cannabis in medically ill participants.

The overall goal of this study is to compare active high cannabidiol (CBD)/ low (-)-trans-Δ9- tetrahydrocannabinol (THC) cannabis vs placebo cannabis in patients with serious medical disorders. Participants will be referred from clinicians and will come to the laboratory daily (3-5 times weekly) for cannabis (15.76% CBD; 3.11% Δ-9-THC) vs placebo (0.0% CBD/ 0.01% Δ-9-THC). The cannabis will be vaporized or smoked as a cannabis cigarette. The participants can choose which option they prefer. The cross-over design will be used where participants receive 2 weeks of active cannabis vs two weeks of placebo in counterbalanced order, with participants blinded to the condition. The outcome measures primarily include measures of pain, with secondary measures of mood, nausea/appetite, quality of life, and the both the potentially positive and negative subjective effects of cannabis (e.g., high, mellow, anxious, paranoid).

ELIGIBILITY:
Inclusion Criteria:

1. One of the medical diagnoses (cancer, amyotrophic lateral sclerosis, Parkinson's disease, spinal cord injury, neuropathy, and phantom limb pain, thalamic pain, pain related to injury of nerve plexus/plexi, and neuropathic facial pain), with reports of pain (at least 3 on item 3 on the 9 item Brief Pain Inventory)that remains despite their current medical treatment.
2. Age 21-60
3. Able to give informed consent, and comply with study procedures
4. Experience inhaling substances.

Exclusion Criteria:

1. Meet DSM-V criteria for current major psychiatric illness, such as bipolar disorder, major depression, active suicidality, or psychosis, that could be exacerbated by the administration of cannabis
2. Meet criteria for major neurological disorder, such as mild cognitive impairment or neurodegenerative disorders (such as movement disorders, dementia), that could be exacerbated by the administration of cannabis.
3. Women who are not practicing an effective form of birth control (condoms, diaphragm, birth control pill, IUD) or currently pregnant
4. Current (weekly) use of cannabis
5. Participants on supplemental oxygen
6. Participants with a substance use disorder involving marijuana or opioids.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-28 (Estimated)

PRIMARY OUTCOMES:
Change in pain ratings using the McGill Pain Questionnaire | 4 weeks
  Participants will be asked to rate their pain over the 4 weeks of receiving active cannabis vs placebo.
Change in sickness-related impairment using the Sickness Impact Profile | 4 weeks
  Participants will be asked to rate physical symptoms for the 4 weeks of the study.
changes in physical and emotional well being using the RAND-36 item medical outcomes survey, a health-related quality of life survey instrument | 4 weeks
  RAND-36 item medical outcomes survey taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions.
Changes in symptoms of pain using the 9 item Brief Pain Inventory | 4 weeks

SECONDARY OUTCOMES:
Change in cognitive status using the Short Portable Mental Status Questionnaire (SPMSQ) | 4 weeks
Change in symptom prevalence, characteristics and degree of stress using the Memorial Symptom Assessment Scale (MSAS) | 4 weeks
Change in the psychological state and psychological well being using the Mental Health Inventory-5 (MHI-5) | 4 weeks
Changes in quality of life using the Multidimensional Index of Life Quality (MILQ) Questionnaire | 4 weeks
Changes in quality of life using the McGill Quality of Life Questionnaire | 4 weeks
Change in symptoms of pain, mood and appetite using the Edmonton Symptom Assessment System (ESAS) | 4 weeks
Memorial Symptom Assessment Scale (MSAS) | 4 weeks
Change in mood using the Hamilton Depression Rating Scale | 4 weeks
Change in mood Hamilton Anxiety Rating Scale | 4 weeks
Change in mood using the Montgomery-Asberg Depression Rating Scale | 4 weeks
Change in mood and quality of life using the Columbia Suicide Severity Rating Scale | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Diana Martinez, MD, Principal Investigator — New York Sate Psychiatric Institute/ Columbia University

IPD SHARING:
Plan to Share IPD: No